CLINICAL TRIAL: NCT05412511
Title: Metabolic Cost of Medicine Ball Training
Acronym: MΒT-UTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MΒT-UTH
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Body Composition; Physical Fitness; Energy Expenditure; Resting Metabolic Rate
Keywords: functional fitness training; Medicine ball Training; Energy Expenditure; Oxygen Consumption; Resistance Trianing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Participants in this arm will perform seven medicine ball training exercises (acute bout per exercise) at two different conditions [Throwing a ball (TB) and no Throwing a ball (NTB)].
  Interventions: Behavioral: MB-TB; Behavioral: MB-NTB
- Control (No Intervention): Participants in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: MB-TB — Training exercises with throwing a medicine ball will be performed for 30 seconds and the training volume will be consisted of 1 repetition.
  Arms: Training
Behavioral: MB-NTB — Training exercises without throwing a medicine ball will be performed for 30 seconds and the training volume will be consisted of 1 repetition.
  Arms: Training

SUMMARY:
In this study, the investigators will be able to estimate the metabolic cost of several foundational medicine ball training exercises.

DETAILED DESCRIPTION:
Medicine ball training has become a popular cardiovascular training choice in fitness centers and athletic performance enhancement facilities. Despite widespread use and growing popularity, little is known about the metabolic demands of such a training method. Therefore, the purpose of this study was to quantify the cardiovascular and metabolic cost from various foundational medicine ball exercises in order to contribute to a better planning of exercise programs in the real world.

Ten healthy young adults were assigned to execute fourteen bodyweight exercises (acute bout) of which seven exercises will be executed by throwing the medicine ball and seven exercises will be executed without a medicine ball throw. Anthropometric, metabolic, functional capacity and performance measurements were conducted at baseline. The metabolic cost was estimated from heart rate, blood lactate, resting oxygen uptake, exercise oxygen uptake, and excess post-exercise oxygen consumption measurements using a portable gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years
* Physically active individuals
* Free of chronic diseases
* Free of musculoskeletal injuries
* Nonsmokers

Exclusion Criteria:

* Musculoskeletal injuries
* Chronic diseases
* Use of alcohol, caffeine and any type of ergogenic supplements or medication before (≤6 months) and throughout the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in exercise-induced energy expenditure | At pre-exercise, during, and 30 minutes after the exercise session (a single bout lasting 30 seconds)
  Exercise energy expenditure (kcal) will be measured using a portable indirect calorimetry system
Change in excess post-exercise oxygen consumption (EPOC) | At 1 hour after exercise session (single bout lasting 30 seconds)
  EPOC (kcal) will be measured using a portable indirect calorimetry system
Change in blood lactate concentration (BLa) | At pre-exercise and 3 minutes after exercise session (a single bout lasting 30 seconds)
  BLa (mmol/L) concentration will be measured in a microphotometer with commercially available kits.
Change in heart rate | At pre-exercise, during, and 30 minutes after ther exercise session (a single bout lasting 30 seconds)
  Heart rate (bpm) will be measured with a wearable heart rate monitor
Change in perceived exertion | At pre-exercise, during, and 30 minutes after the exercise session (a single bout lasting 30 seconds)
  Rating of perceived exertion (RPE) will be measured with the Borg scale (0-10)

SECONDARY OUTCOMES:
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | At baseline
  BMI will be calculated using the Quetelet's equation
Waist circumference (WC) | At baseline
  WC (cm) will be measured using a Gullick II tape
Hip circumference (HC) | At baseline
  HC (cm) will be measured using a Gullick II tape
Waist-to-hip ratio (WHR | At baseline
  WHR will be calculated by dividing the waist by the hip measurement
Resting metabolic rate (RMR) | At baseline
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Body fat (BF) Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA) | At baseline
  BF (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass (FM)t Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA) | At baseline
  FM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat-free mass (FFM) | At baseline
  FFM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Maximal oxygen consumption (VO2max) | At baseline
  VO2max (mL/kg/min) will be assessed by a portable open-circuit spirometry system
Maximal strength (1RM) | At baseline
  1RM (kg) will be measured bilaterally on a horizontal leg press and seated chest press machine.
Muscular endurance | At baseline
  Muscular endurance (repetitions) will be measured on a 1-min curl-up and push-up test.
Functional capacity | At baseline
  Functional capacity will be assessed using a movement-based screening tool titled Functional Movement Screening (FMS). The FMS will be consisted of 7 movement tasks that will be scored from 0 to 3 points and the sum will create score ranging from 0 to 21 points (0 = pain with pattern regardless of quality, 1 = unable to perform pattern, 2 = able to perform pattern with compensation/imperfection, 3 = able to perform pattern as directed)Functional capacity will be assessed using a movement-based screening tool titled Functional Movement Screening (FMS). The FMS will be consisted of 7 movement tasks that will be scored from 0 to 3 points and the sum will create score ranging from 0 to 21 points (0 = pain with pattern regardless of quality, 1 = unable to perform pattern, 2 = able to perform pattern with compensation/imperfection, 3 = able to perform pattern as directed)

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Study Director — University of Thessaly
Locations (1):
- Laboratory of Exercise Physiology, Exercise Biochemistry and Sports Nutrition, School of Physical Education, Sports Sciences and Dietetics, University of Thessaly, Trikala, Greece